CLINICAL TRIAL: NCT04585308
Title: Prospective, Multi-center, Single-Arm Feasibility Study of the transShield Embolic Protection System
Brief Title: transShield Embolic Protection System Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransAortic Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-05-001
Record Dates: First submitted 2020-10-05; First posted 2020-10-14 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm (Experimental): Patients with severe native aortic valve stenosis who meet the commercially approved indications for TAVR.
  Interventions: Device: transShield Embolic Protection System

INTERVENTIONS:
Device: transShield Embolic Protection System — Used for embolic protection during TAVR.

SUMMARY:
The objective of this study is to evaluate the safety and performance of the transShield Embolic Protection System (EPS) used for embolic protection during Transcatheter Aortic Valve Replacement (TAVR).

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm feasibility study to assess the safety and performance of the transShield EPS. Patients with severe native aortic valve stenosis scheduled for TAVR will be screened for study eligibility. Subjects who meet the commercially approved indications for TAVR and comply with the study inclusion/exclusion criteria are eligible for enrollment. Patients will be followed for 30 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria to be eligible for participation in the study:

  * Patient is >18 years old
  * Patient is scheduled for percutaneous TAVR with up to 20French compatible commercial TAVR system
  * Patient meets indications for TAVR per the device Instructions For Use
  * The diameter of the artery at the site of the filter placement is between 28 mm and 42 mm
  * Size and condition of the femoral artery iliac arteries are appropriate for the 12French transShield Expandable Introducer and 20F Embolic Protection Device
  * Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated procedures
  * Patient is willing and able to complete follow-up requirements

Exclusion Criteria:

* Patients must be EXCLUDED from participation in this study if any of the following criteria are met:

  * Patient not undergoing TAVR via the trans-femoral route
  * Carotid artery stenosis >70% in either carotid artery
  * Severe vascular tortuosity or anatomy that would preclude the safe introduction of the device
  * Aortic valve is a congenital unicuspid or congenital bicuspid valve or is non-calcified
  * Mixed aortic valve disease (aortic stenosis and aortic regurgitation with predominant aortic regurgitation >3+)
  * A known contraindication or hypersensitivity to all anticoagulation regimens or an inability to undergo anticoagulation for the study procedure
  * History of bleeding diathesis or in whom anticoagulant and/or anti-platelet therapy is contraindicated, patients who will refuse transfusion, or havean active peptic ulcer or upper GI bleeding within the prior 3 months
  * Renal insufficiency, defined as a creatinine level > 221μmol/L and/or end-stage renal disease requiring chronic dialysis at time of treatment
  * History of stroke or transient ischemic attack (TIA) within prior 6 months
  * Evidence of an acute myocardial infarction (MI) within prior 30 days
  * Hemodynamic or respiratory instability requiring inotropic support, mechanical ventilation, or mechanical heart assistance within prior 30 days
  * Hypertrophic cardiomyopathy with or without obstruction
  * Need for emergency surgery for any reason
  * Severe left ventricular (LV) dysfunction with LV ejection fraction (LVEF) <20%
  * Severe pulmonary hypertension and right ventricular (RV) dysfunction
  * Echocardiographic evidence of intracardiac mass, thrombus or vegetation
  * Life expectancy < 12 months due to non-cardiac co-morbid conditions
  * Evidence of active systemic or local groin infection
  * Significant aortic disease, including abdominal aortic or thoracic aneurysm defined as maximal luminal diameter 5cm or greater; marked tortuosity (hyperacute bend), aortic arch atheroma or narrowing (especially with calcification and surface irregularities) of the abdominal or thoracic aorta, severe "unfolding" and tortuosity of the thoracic aorta
  * Known hypersensitivity or contraindication to aspirin, heparin, ticlopidine, or clopidogrel, or sensitivity to contrast media, that cannot be managed with premedication
  * Planned other cardiac surgical procedure within 2 weeks prior to, or planned cardiac surgical or interventional procedure within 30 days after the TAVR procedure. Note: Diagnostic cardiac catheterization is permitted within 10 days prior to the TAVR procedure
  * Neurodegenerative or other progressive neurological disease
  * Known allergy to any device component
  * Known or suspected to be pregnant or lactating
  * Currently enrolled in an investigational drug or device clinical study in which the primary endpoint has not occurred
  * Patient has other medical, social or psychological problem that in the opinion of the investigator precludes them from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Safety - Incidence of 30-Day combined rate of the following events directly related to the transShield EPS as defined by VARC-2 | 30 day combined rate post-procedure
  * Major Adverse Cardiac and Cerebrovascular Events (MACCE)
    * All cause mortality
    * All cause stroke (disabling and non-disabling)
    * Acute kidney injury (Stage 2 or 3)
  * Major vascular complications
Performance - Technical Success defined as the transShield EPS ability to perform all the following functions without adjudicated device malfunction | During the procedure
  * Ability to successfully deploy the device in the correct anatomical position, in the ascending aorta without interference with TAVR procedure/devices
  * Ability to retrieve and remove the device intact, including no visual evidence of any filter damage

SECONDARY OUTCOMES:
Safety - Incidence of minor vascular complications directly related to the transShield EPS as defined by VARC-2. | 30 days post-procedure
  * As defined by VARC-2.
  * Incidence of peri-procedural disabling stroke as defined by a modified Rankin Scale (mRS) score of 2 or more at 30 days and an increase in at least one mRS category from an individual's pre-stroke baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Webster, MD, Principal Investigator — Auckland City Hospital; Carlos Calderas, MD, Principal Investigator — Policlinica Metropolitana - Venezuela
Locations (4):
- New Zealand (2):
  - Auckland City Hospital, Auckland, Grafton
  - Waikato Hospital, Hamilton
- Venezuela (2):
  - Policlinica Metropolitana, C.A, Miranda, Miranda
  - Ascardio Asociación Cardiovascular Centroccidental, La Lara, Sector La Feria

IPD SHARING:
Plan to Share IPD: No